CLINICAL TRIAL: NCT04096846
Title: Relationship Between Vitamin D Deficiency and Oral Mucositis in Patients With Acute Lymphoblastic Leukemia Receiving Methotrexate in South Egypt Cancer Institute , a Prospective Study
Brief Title: Effect of Vitamin D Diffiency on Oral Mucosa in Patients Recieving Methotrexate Chemotherapy
Acronym: VitDandMTX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magy Ibrahim Anis Rizkallah, Demonstrator of cancer biology, Assiut University
Other Study IDs: Vit D and oral mucositis
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laboratory investigation — detection of serum level of methotrexate and serum level of vitamin D

SUMMARY:
it's a prospective study aiming to improve quality of life of patients with acute lymphoblastic leukemia suffering from oral mucositis, receiving courses of methotrexate chemotherapy , by measuring vitamin D in those patients before induction therapy and the change in its level during treatment, that associated with methotrexate-induced oral mucositis, taking in consideration serum level of methotrexate, so we may have assiotiation between vitamin D difficiency and oral mucositis . at the end we can have preventive interventions to protect against this harmful side effect.

DETAILED DESCRIPTION:
Treatment outcome of acute lymphoblastic leukemia (ALL) is improved recently and the 5-year survival rates reached 90% in developed countries . So more research currently focuses on strategies to decrease toxic adverse effects of methotrexate (MTX). Oral mucositis occurs in about 20% of patients receiving methotrexate Identifying risk factors leading to this side effects would be valuable to develop preventive interventions and improve quality of life for these patients .

Previous studies revealed a relationship between vitamin D deficiency and chemotherapy-induced oral mucositis in cancer patients. This hormone is important in many physiological processes in the body as bone mineralization and immune regulations. The main sourses of Vitamin D is production in the skin through sunlight exposure, diet and Vitamin D supplements .

Previous literature showed that receptors for vitamin D expressed in the mucosa and so there is a relationship between vitamin D deficiency and increase inflammation and impairment of mucosa .

Patients with acute lymphoblastic leukemia maybe at risk of vitamin D deficiency because of impaired vitamin intake and sunlight exposure . In this study we examin the possible role of vitamin D in relation to methotrexate induced oral mucositis in cancer patients.

* peripheral blood samples from patients before starting chemotherapy course with methotrexate and 24 hr after starting the treatment for measurement level of vitamin D, samples centrifuged at the speed of 2000 - 3000 rpm for 20 min , then analyzed using ELISA.
* blood samples after treatment also used to determine serum level of methotrexate which may lead to toxic adverse effect as oral mucositis , samples centrifuged at speed of 2000 - 3000 rpm for 10 min and analyzed using Viva-E equipment.
* All serum samples were stored at -80 °C and analyzed collectively

ELIGIBILITY:
Inclusion Criteria:

* patients with acute lymphocytic leukemia in South Egypt Cancer Institute
* patients recieving methotrexate in protocol of treatment
* both sex included

Exclusion Criteria:

* patients with other types of tumors
* patients refuse to join the research
* patients with comorbid hepatic or renal impairment

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric and old patients with acute lymphocytic leukemia treated with methotrexate based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Relation between vitamin D difficiency and oral mucositis in patients with leukemia | baseline 6 months to 1 year
  Difficiency of vitamin D in patients with acute lymphoblastic leukemia recieving methotrexte assiociated with oral mucositis and so later on we can improve thier quality of life by supplying vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Mahmoud Hamdy, Phd, Study Director — Assiut University; Nevin Abdelazim Abelalim, Phd, Study Director — Assiut University

REFERENCES:
- [Background] Al-Maweri SA, Halboub E, Al-Sufyani G, Alqutaibi AY, Shamala A, Alsalhani A. Is vitamin D deficiency a risk factor for recurrent aphthous stomatitis? A systematic review and meta-analysis. Oral Dis. 2020 Sep;26(6):1116-1123. doi: 10.1111/odi.13189. Epub 2019 Oct 8. PMID 31493304
- [Background] Anand A, Singh S, Sonkar AA, Husain N, Singh KR, Singh S, Kushwaha JK. Expression of vitamin D receptor and vitamin D status in patients with oral neoplasms and effect of vitamin D supplementation on quality of life in advanced cancer treatment. Contemp Oncol (Pozn). 2017;21(2):145-151. doi: 10.5114/wo.2017.68623. Epub 2017 Jun 30. PMID 28947884
- [Background] Oosterom N, Dirks NF, Heil SG, de Jonge R, Tissing WJE, Pieters R, van den Heuvel-Eibrink MM, Heijboer AC, Pluijm SMF. A decrease in vitamin D levels is associated with methotrexate-induced oral mucositis in children with acute lymphoblastic leukemia. Support Care Cancer. 2019 Jan;27(1):183-190. doi: 10.1007/s00520-018-4312-0. Epub 2018 Jun 19. PMID 29922939
- [Background] Lalla RV, Choquette LE, Feinn RS, Zawistowski H, Latortue MC, Kelly ET, Baccaglini L. Multivitamin therapy for recurrent aphthous stomatitis: a randomized, double-masked, placebo-controlled trial. J Am Dent Assoc. 2012 Apr;143(4):370-6. doi: 10.14219/jada.archive.2012.0179. PMID 22467697